CLINICAL TRIAL: NCT02181478
Title: Intra-osseous Co-transplant of Cord Blood and Mesenchymal Stromal Cells: A Feasibility Study
Brief Title: Intra-Osseous Co-Transplant of UCB and hMSC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marcos de Lima, Principal Investigator, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1Z14; NCI-2014-01316 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE1Z14 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndromes; Myelofibrosis; Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Relapsed Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Lymphoid Malignancies; Chronic Myelogenous Leukemia
Keywords: Total Body Irradiation; Human Mesenchymal Stromal Cells; hMSC; Cyclophosphamide; Fludarabine; Dimethyl Sulfoxide; DMSO; Cyclosporine; Mycophenolate Mofetil; MMF; Granulocyte- Colony Stimulating Factor; G-CSF; GVHD; Cancer; feasibility
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Primary Myelofibrosis; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms | interventions — Cyclophosphamide; fludarabine phosphate; Whole-Body Irradiation; Cyclosporine; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Transplantation; Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (intra-osseous UCB with hMSC co-transplant) (Experimental): REDUCED INTENSITY CONDITIONING (RIC):
  Flu/Cy/TBI: Patients receive cyclophosphamide IV over 2 hours on day -6 and fludarabine phosphate IV on days -6 to -2 and undergo total-body irradiation on day -1.
  Flu/Mel: Patients receive fludarabine daily on days -5 to -2, a single dose of melphalan on day -2, and ATG on day -3 and day-2.
  GVHD PROPHYLAXIS: Patients receive cyclosporine PO or IV over 2 hours every 12 hours on beginning on days -5 to 100 with taper beginning on day 100 and mycophenolate mofetil IV or PO BID on days -5 to 100.
  TRANSPLANT: Patients undergo a co-transplantation of an intra-osseous umbilical cord blood transplantation and a mesenchymal stem cell transplantation on day 0.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Radiation: total-body irradiation; Drug: cyclosporine; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Procedure: mesenchymal stem cell transplantation

INTERVENTIONS:
Drug: cyclophosphamide — All patients will receive a single IV dose of 50 mg/kg of cyclophosphamide on day -6
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: fludarabine phosphate — Given by IV during prep at 40mg/m2 for 5 days
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Undergo single fraction of reduced intensity conditioning (RIC) regimen of 200 cGy TBI without shielding on day -1
  Other Names: TBI
Drug: cyclosporine — Initiated in patients on the day -5. Cyclosporine will be administered orally or intravenously at 2 mg/kg/dose every 12 hours for 2-hour period. Cyclosporine will continue until day +100
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given at 1g intravenously or orally twice daily from day -5 to +100, or as clinically indicated.
  Other Names: Cellcept; MMF
Procedure: umbilical cord blood transplantation — Following RIC, on day T+0, dimethylsulphoxide will be removed from the cord blood cells and given as transplant.
  Other Names: cord blood transplantation; transplantation, umbilical cord blood; UCB transplantation
Procedure: mesenchymal stem cell transplantation — The total dosage of hMSC will be 2x10^6cells/kg (+/-20%).
  Other Names: hMSC transplantation

SUMMARY:
This clinical trial studies intra-osseous donor umbilical cord blood and mesenchymal stromal cell co-transplant in treating patients with hematologic malignancies. Giving low doses of chemotherapy and total-body irradiation before a co-transplant of donor umbilical cord blood and mesenchymal stromal cells into the bone (intra-osseous) helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil at the time of transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the feasibility of combining intra-osseous umbilical cord blood (UCB) hematopoietic stem cells and human mesenchymal stromal cells (hMSC) following reduced intensity conditioning (RIC).

SECONDARY OBJECTIVES:

I. To estimate the time to engraftment of intra-osseous (IO) UCB transplant combined with hMSC following RIC.

II. To estimate the safety profile of IO UBC transplant combined with hMSC.

OUTLINE:

REDUCED INTENSITY CONDITIONING: Patients receive cyclophosphamide intravenously (IV) over 2 hours on day -6 and fludarabine phosphate IV on days -6 to -2 and undergo total body irradiation (TBI) on day -1.

GRAFT-VERSUS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive cyclosporine orally (PO) or IV over 2 hours every 12 hours on beginning on days -5 to 100 with taper beginning on day 100 and mycophenolate mofetil IV or PO twice daily (BID) on days -5 to 100.

TRANSPLANT: Patients undergo intra-osseous UCB and hMSC co-transplant on day 0.

After completion of study treatment, patients are followed up at days 28 and 100, and then at 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following malignancies:

  * Acute myelogenous leukemia (AML): high-risk AML including:

    * Antecedent hematological disease (e.g., myelodysplasia [MDS])
    * Treatment-related leukemia
    * Complete remission (first complete remission [CR1]) with poor-risk cytogenetics or molecular markers (e.g. fms-related tyrosine kinase 3 [Flt 3] mutation, 11q23, del 5, del 7, complex cytogenetics)
    * Second complete remission (CR2) or third complete remission (CR3)
    * Induction failure or first relapse with either

      * ≤ 10% blasts in the marrow and/or
      * ≤ 5% blasts in the peripheral blood
  * Acute lymphoblastic leukemia (ALL)

    * High-risk CR1 including:
    * Poor-risk cytogenetics (e.g., Philadelphia chromosome t(9;22)or 11q23 rearrangements)
    * Presence of minimal disease by flow cytometry after 2 or more cycles of chemotherapy
    * No complete remission (CR) within 4 weeks of initial treatment
    * Induction failure
    * CR2 or CR3 with either:

      * ≤ 10% blasts in the marrow and/or
      * ≤ 5% blasts in the peripheral blood
  * Myelodysplastic syndromes (MDS), Intermediate-1 (INT-1), intermediate-2 (INT-2) or high Revised International Prognostic Scoring System (IPSS-R) score that has failed at least 1 first line therapy
  * Myelofibrosis (MF):

    * Intermediate-2 or high risk by Dynamic International Prognostic Scoring System (DIPSS)-plus
    * Monosomal karyotype
    * Presence of inv(3)/i(17q) abnormalities
    * Other unfavorable karyotype OR leukocytes ≥40 X 10^9/L AND
    * Circulating blasts ≤ 9%
  * Relapsed or refractory lymphoid malignancies (including non-Hodgkin lymphoma, Hodgkin lymphoma and chronic lymphocytic leukemia) meeting the following criteria:

    * Disease status: stable disease, partial remission or 2nd and 3rd complete remission
  * Chronic myelogenous leukemia (CML) in second chronic phase after accelerated or blast crisis; blast crisis defined as:

    * Blast count ≥ 20% in the peripheral blood or bone marrow
    * Large foci of blasts on bone marrow
    * Presence of extra-medullary blastic infiltrate (myeloid sarcoma or chloroma)
  * Recipients of prior autologous or allogeneic transplant are eligible, as long as at least 3 months have passed since the transplant, and the patient fulfills other eligibility criteria
  * Eastern Cooperative Oncology Group (ECOG) performance status ≤2
  * Candidates for reduced intensity conditioning regimens
  * Patients who do not have HLA-matched (defined as matched in HLA A, B, C, and DRB1) related or unrelated donors, those who elect to undergo UCB even if they have a MRD or MUD, or patients who require a UCB either for emergency indications such as primary graft failure.
  * Cord Blood Units available through NMDP with the following minimal criteria:

    * HLA Match: 4/6 or better match (HLA A, B, DRB1)
    * Cell dose: Minimum of 2.0x107TNC/kg pre thaw
  * Concurrent therapy for extramedullary leukemia or central nervous system (CNS) lymphoma: concurrent therapy or prophylaxis for testicular leukemia, CNS leukemia, and CNS lymphoma including standard intrathecal chemotherapy and/or radiation therapy will be allowed as clinically indicated; such treatment may continue until the planned course is completed; subjects must be in CNS remission at the time of protocol enrollment if there is a history of CNS involvement
  * Subjects must have a back-up umbilical cord on the registry in addition to the umbilical cord being used in this study
  * Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with inadequate Organ Function as defined by:

  * Creatinine clearance < 30 ml/min
  * Bilirubin ≥ 2 x institutional upper limit of normal
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≥ 2 x institutional upper limit of normal
  * Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≥ 2 x institutional upper limit of normal
  * Corrected diffusing capacity of the lung for carbon monoxide (DLCOcorr) < 40% normal
* Left ventricular ejection fraction < 35%
* Patients with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women are excluded from this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with BM cellularity failure: Measure of feasibility | 42 days after transplant
  Primary graft failure is defined by <10% BM cellularity in bone marrow biopsies. Failure in more than 30% of patients will indicate unfeasibility of treatment
Number of patients with ANC failure without evidence of disease: Measure of feasibility | 42 days after transplant
  Primary graft failure is defined by <500 ANC cell/ul in bone marrow biopsies. Failure in more than 30% of patients will indicate unfeasibility of treatment
Number of patients with hematopoietic recovery without evidence of donor umbilical cord blood engraftment: Measure of feasibility | 42 days after transplant
  Primary graft failure is defined by hematopoietic recovery with <10% donor cell chimerism. Failure in more than 30% of patients will indicate unfeasibility of treatment
Number of patients with hematopoietic recovery without evidence of donor umbilical cord blood engraftment: Measure of feasibility | 100 days after transplant
  Primary graft failure is defined by hematopoietic recovery with <40% donor cell chimerism. Failure in more than 30% of patients will indicate unfeasibility of treatment

SECONDARY OUTCOMES:
Incidence of toxicities assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 12 months
  Descriptive statistics will be used.
Rate of neutrophil recovery | Up to 12 months
  The rate of neutrophil recovery and median time of recovery will be estimated using the methods of Kaplan and Meier.
Rate of platelet recovery | Up to 12 months
  The rate of platelet recovery and median time of recovery will be estimated using the methods of Kaplan and Meier.
Median time of neutrophil recovery | Up to 12 months
  The median time of neutrophil recovery will be estimated using the methods of Kaplan and Meier.
Median time of platelet recovery | Up to 12 months
  The median time of platelet recovery will be estimated using the methods of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States